CLINICAL TRIAL: NCT05215496
Title: [18F]Fluoro-PEG-folate PET/CT Imaging in Epithelial Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Reached the stop criteria after the interim analysis
Sponsor: Lioe-Fee de Geus-Oei, MD PhD (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Centre for Human Drug Research, Netherlands (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Lioe-Fee de Geus-Oei, MD PhD, Principal Investigator, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P20.048; 2020-000112-29 (EudraCT Number); NL72618.058.20 (Other: Medical ethical committee Leiden Den Haag Delft)
Record Dates: First submitted 2021-09-01; First posted 2022-01-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: 185 MBq of [18F]fluoro-PEG-folate PET tracer will be intravenously administered to 15 patients with radiologically advanced stage EOC who are scheduled to undergo cytoreductive surgery, after which an FR-targeted PET/CT will be made. FR-targeted PET/Ct results will be compared to the intraoperative findings, postoperative histopathology (gold standard) and the conventional CT scan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F]fluoro-PEG-folate PET/CT scan (Experimental): Patients with FIGO stage IIIB/IIIC epithelial ovarian cancer, 185 MBq of [18F]fluoro-PEG-folate.
  Interventions: Diagnostic Test: [18F]fluoro-PEG-folate PET/CT scan

INTERVENTIONS:
Diagnostic Test: [18F]fluoro-PEG-folate PET/CT scan — A dynamic FR-targeted PET scan, a low-dose CT scan without contrast agents, and a static FR-targeted PET scan will be obtained

SUMMARY:
The pre-operative assessment of intra-abdominal tumor load in patients with epithelial ovarian cancer (EOC) remains unreliable with standard imaging modalities. The use of tumor targeted imaging, such as folate receptor (FR)-targeted positron emission tomography (PET) imaging could aid in the preoperative assessment of metastatic tumor load.

This study aims to evaluate the safety and tolerability, and pharmacokinetics of the [18F]fluoro-PEG-folate PET tracer and to assess the sensitivity and specificity of a [18F]fluoro-PEG-folate PET/CT scan for the preoperative detection of intra-abdominal metastatic lesions in patients with advanced stage epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients with radiologically FIGO stage IIIB/IIIC EOC based on the conventional CT scan who are:

* scheduled to undergo primary cytoreductive surgery and

  1. in whom EOC is histologically proven, or
  2. in whom EOC is cytologically suspected and a serum CA125/CEA ratio > 25 is found

or

* treated with neoadjuvant chemotherapy (NACT) and are scheduled to undergo interval cytoreductive surgery and

  1. in whom EOC is histologically proven, or
  2. in whom EOC is cytologically suspected and a serum CA125/CEA ratio > 25 was found before NACT
  3. and with radiologically FIGO stage IIIB/IIIC EOC based on the response evaluation CT scan after NACT

Exclusion Criteria:

1. Women younger than 30 years of age (in accordance with the guidelines of the Netherlands Commission on Radiation Dosimetry [23], as the total radiation dose will be 7.2 mSv)
2. Patients who previously underwent primary laparotomy and in whom complete or optimal cytoreduction was not considered feasible.
3. Contraindication for PET (pregnancy, lactating or severe claustrophobia)
4. Thrombocytopenia (platelet count < 100 x 10^9/L) and/or INR > 2
5. Impaired renal function (defined as eGFR < 50 mL/1.73 m2)
6. Impaired liver function (ALT, AST or total bilirubin > 3x upper limit of normal)
7. Clinically significant abnormalities on ECG and/or clinically laboratory test
8. Inability to tolerate lying supine for the duration of a PET/CT examination (~110 minutes)
9. Patients with concomitant malignancy (except basal cell carcinoma of the skin) or any condition that in the opinion of the investigators could potentially jeopardize the health status of the patient
10. Patients not able to comply with the study procedures
11. Patients who did not give informed consent

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of the [18F]fluoro-PEG-folate PET tracer | From administration up to two hours after administration
  To assess the tolerability of the [18F]fluoro-PEG-folate PET tracer vital signs will be recorded every 15 minutes starting directly before administration and continued up to two hours after dosing. The endpoint for this study is the number of patients whose vital signs stayed within a normal range of their baseline.
Arterial plasma input curve of the [18F]fluoro-PEG-folate tracer | At regular intervals up to 90 minutes post injection of the tracer.
  Blood samples will be collected to determine the arterial plasma input curve of the tracer.
Pharmacokinetic distribution of the [18F]fluoro-PEG-folate tracer | At regular intervals up to 90 minutes post injection of the tracer.
  Blood samples will be collected to determine the pharmacokinetic distribution of the tracer.
Safety of the [18F]fluoro-PEG-folate PET tracer | Up to six weeks after the injection of the tracer.
  Total number of AEs and SAEs that occur during the observation period.

SECONDARY OUTCOMES:
Sensitivity and specificity | Up to 6 weeks after the FR-targeted PET/CT scan.
  Sensitivity and specificity of the FR-targeted PET/CT scan for the detection of metastatic EOC lesions. Postoperative histopathology will serve as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Lioe-Fee de Geus-Oei, MD, PhD, Principal Investigator — LUMC
Locations (1):
- Katja Gaarenstroom, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ciggaar IA, de Muynck LDAN, de Geus-Oei LF, van Velden FHP, de Kroon CD, Pereira Arias-Bouda LM, Noortman WA, van Persijn van Meerten EL, Dibbets-Schneider P, Helmerhorst HJF, Windhorst AD, Vahrmeijer AL, Peters ITA, Gaarenstroom KN. Preoperative [18F]fluoro-PEG-folate PET/CT in advanced stage epithelial ovarian cancer: A safety and feasibility study. Nucl Med Biol. 2024 Nov-Dec;138-139:108952. doi: 10.1016/j.nucmedbio.2024.108952. Epub 2024 Sep 19. PMID 39326323